CLINICAL TRIAL: NCT04812106
Title: Long Chain Fatty Acid Oxidation Disorders (LC-FAOD) Online Disease Monitoring Program (DMP)
Brief Title: Long-Chain Fatty Acid Oxidation Disorders Online Disease Monitoring Program
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision not related to safety concerns
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: UX007-CL402
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Long-chain Fatty Acid Oxidation Disorders (LC-FAOD)
Keywords: CACT Deficiency; Carnitine Acylcarnitine Translocase Deficiency; Long-chain 3-hydroxyacyl-CoA Dehydrogenase Deficiency; TFP Deficiency; Trifunctional Protein Deficiency; CPT1; CPT2; Carnitine Palmitoyltransferase Deficiencies; Very Long Chain Acyl Coa Dehydrogenase Deficiency; VLCAD; LCHAD; CPT I; CPT II
MeSH Terms: conditions — Carnitine-Acylcarnitine Translocase Deficiency; Trifunctional Protein Deficiency With Myopathy And Neuropathy; VLCAD deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with LC-FAOD
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The objectives of this study are to characterize the disease impact, the disease management and resource utilization, and provide benefits to the LC-FAOD community, by use of a convenient online platform for participants (or caregivers) to self-report information.

DETAILED DESCRIPTION:
The online LC-FAOD DMP is a non-interventional, prospective, observational disease-monitoring program conducted through a mobile/web-based application developed by the Sponsor. Participant data will be captured via the mobile/web-based application and entered into the database designed and maintained by the Sponsor and/or its designee. Additional objectives of the study are to benefit the LC-FAOD community by developing a comprehensive database for use by the LC-FAOD community to characterize patient experience, inform disease management, and enable further research, utilize the digital platform to notify patients, caregivers, and relevant patient advocacy groups of research studies and clinical trials and share aggregated and de-identified outputs to facilitate the exchange of information with patients and/or caregivers.

Participants can be on any treatment in order to participate. Medical management of the disease should continue as directed by the patient's physician(s). Specifically, no treatments, investigational agents, or experimental interventions will be provided as part of this online LC-FAOD DMP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of LC-FAOD including: carnitine palmitoyltransferase (CPT I or CPT II) deficiency, very long chain acyl-CoA dehydrogenase (VLCAD) deficiency, long-chain 3-hydroxyacyl-CoA dehydrogenase (LCHAD) deficiency, trifunctional protein (TFP) deficiency, or carnitine-acylcarnitine translocase (CACT) deficiency.
* Willing and able to provide consent or, if a minor, provide assent and informed consent by their legally authorized representative.
* Access to the internet and an internet-enabled device.
* Reside in the geographical regions where the platform is supported and approved by applicable IRB/IEC and /or health authority.
* Not receiving triheptanoin through an Ultragenyx-sponsored interventional clinical trial or Ultragenyx Investigator Sponsored Trial (IST). NOTE: Individuals are eligible to participate in this online DMP if they previously participated in UX007 clinical trials, are currently participating in the in clinic UX007-CL401 (NCT04632953), are receiving triheptanoin through Expanded Access or Compassionate Use programs, or are receiving commercially available triheptanoin via prescription.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The aim of the online LC-FAOD DMP is to enroll a broad spectrum of individuals with confirmed diagnosis of any LC-FAOD type. No limit will be placed on sample size. Individuals of all ages, including caregivers of newborns and minors, are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
LC-FAOD Management: Nutrition and Dosing Utilized to Control LC-FAOD | 10 years
LC-FAOD At-home Interventions: Types of Interventions Used | 10 years
  Interventions used to prevent or mitigate Major Clinical Events (MCEs)
LC-FAOD MCEs: Annualized Event Rate of all MCEs | 10 years
  MCEs include skeletal myopathy (rhabdomyolysis), hepatic (hypoglycemia, liver dysfunction), and cardiac disease (cardiomyopathy) events. An MCE is defined as any visit to the ED/acute care, hospitalization, emergency intervention (ie, any unscheduled administration of therapeutics in the clinic), or any similar event whether caused primarily by LC-FAOD or by an intercurrent illness complicated by LC-FAOD
LC-FAOD MCEs: Annualized Event Days in the Emergency Department (ED)/Hospital for all MCEs | 10 years
LC-FAOD MCEs: Time to First MCE in all Newborn Patients (<=1 Year) | 10 years
Disease Management as Assessed by Physical Activity | 10 years
Patient Reported Outcomes: Infant and Toddler Quality of Life Questionnaire (ITQOL) Short Form | 10 years
Patient Reported Outcomes: Short-Form 10 (SF-10) Health Survey for Children | 10 years
Patient Reported Outcomes: Medical Outcomes Study 12-Item Short Form Version 2 (SF-12v2) for Adults | 10 years
Participant Survey: Patient and Caregiver-Reported Outcomes | 10 years
Participant Survey: Disease Symptoms | 10 years
Participant Survey: Schooling and Work Status | 10 years
Participant Survey: Absenteeism/Presenteeism | 10 years
Participant Survey: EuroQol Group 5-dimension 5-level (EQ-5D-5L) Instrument | 10 years
Healthcare Resource Utilization: LC-FAOD-related Medical Resource Use Over Time | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: Ultragenyx Patient Advocacy/LC-FAOD Disease Information — https://ultrarareadvocacy.com/conditions-we-study/long-chain-fatty-acid-oxidation-disorders-lc-faod/